CLINICAL TRIAL: NCT00816348
Title: Compassionate Use of Omegaven IV Fat Emulsion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cindy Haller (Other)
Responsible Party: Sponsor-Investigator, Cindy Haller, Physician, Northwell Health
Organization: Northwell Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-204
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Cholestasis; Total Parenteral Nutrition-induced Cholestasis
Keywords: Cholestasis; Parenteral Nutrition Associated Liver Disease
MeSH Terms: conditions — Cholestasis | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omegaven (Other): All subjects will receive Omegaven
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — Omegaven® will be initiated at a dose of 0.5 gram/kg/day and is infused over 24 hours for 1-2 days, and then advanced to 1 gram/kg/day. Omegaven® will be infused intravenously through either a central or peripheral catheter alone or in conjunction with parenteral nutrition. Omegaven® will continue until weaned from PN. Monotherapy with Omegaven® can continue as an additional source of calories after the dextrose/protein portion of PN is discontinued. Omegaven may be restarted within seven days of discontinuing therapy. After seven days, and meeting inclusion criteria, Omegaven can resume at the initial dose of 0.5 grams/kg/day, advancing to 1 gm/kg/day.

SUMMARY:
This is a compassionate use protocol to use intravenous fish oil infusion, Omegaven®, to infants and children with parenteral nutrition-associated liver disease to enable reversal of elevated serum liver enzymes and direct bilirubin (cholestasis).

DETAILED DESCRIPTION:
Intravenous lipids are necessary in PN (parenteral nutrition) dependent patients due to their high caloric value and essential fatty acid content. However, parenteral fat emulsions composed of soybean oils (omega 6 fatty acids) have been implicated in predisposing patients to PN associated liver disease.

It is hypothesized that by administering Omegaven®, comprised of fish oil (omega 3 fatty acids) in place of conventional soybean fat emulsion, the progression of PN-associated cholestasis may be prevented or reversed.

ELIGIBILITY:
Inclusion Criteria:

* Two consecutive direct bilirubin levels of 2 mg/dl or more in a parenteral nutrition dependent infant or child (unable to meet nutritional needs solely by enteral nutrition)
* Other causes of liver disease have been excluded. A liver biopsy is not necessary for treatment.
* The patient must have utilized standard therapies to prevent the progression of the liver disease including reduction/removal of copper and manganese from daily PN, trial of enteral feeding if possible, and the use of ursodiol (i.e., Actigall®).

Exclusion Criteria:

* Documented causes of chronic liver disease other than parenteral nutrition associated liver disease
* Proven severe advanced liver disease including cirrhosis on biopsy, varices, ascites.
* An allergy to any seafood product, egg protein, and/or previous allergy to Omegaven®
* Active coagulopathy characterized by ongoing bleeding or by a requirement for clotting factor replacement (e.g. fresh frozen plasma or cryoprecipitate) to maintain homeostasis
* Impaired lipid metabolism or severe hyperlipidemia with or without pancreatitis
* Unstable diabetes mellitus or hyperglycemia
* Stroke, embolism, collapse and shock, recent MI
* Cholestasis due to any reason other than parenteral associated liver disease
* Active new infection at time of initiation of Omegaven®
* Hemodynamic instability
* The patient may not be enrolled in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team).

Ages: 2 Weeks to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Haller, MD, Principal Investigator — Cohen Children's Medical Center of New York
Locations (2):
- United States (2):
  - Cohen Children's Medical Cenetr of New York at North Shore, Manhasset, New York
  - Cohen Children's Medical Center of New York, New Hyde Park, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omegaven
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Omegaven
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: days] | 89.3 [35 to 306]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 15
bilirubin level [Mean (Standard Deviation); unit: mg/dL] | 6.79 (4.14)

OUTCOME MEASURES:

1. Primary Outcome: Level of Bilirubin
Description: measurement of bilirubin level weekly. Available data reported.
Time Frame: week 2, 3,4,and 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Omegaven
Number analyzed (Participants) | 15
mg/dL
  Week 2 N=12 | 7.4 (4.38)
  Week 3 N=8 | 6.63 (4.39)
  Week 4 N=10 | 7.97 (6.5)
  Week 8 N=11 | 4.72 (4.81)

ADVERSE EVENTS:
Arm/Group | Omegaven
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omegaven (N=15)
death (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes